CLINICAL TRIAL: NCT04801186
Title: REMPRO Registry A Multi-country, Multi-centre, Non-interventional, Retrospective Study to Describe the Real-world Treatment Patterns and Associated Clinical Outcomes in Patients With Metastatic Castration-resistant Prostates Cancer
Brief Title: Retrospective Study to Describe the Real-world Treatment Patterns and Associated Clinical Outcomes in Patients With Metastatic Castration-resistant Prostates Cancer
Acronym: REMPRO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00037
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Castration-resistant Prostates Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

SUMMARY:
This is a multi-country, multi-centre, retrospective, non-interventional cohort study planned to include patients diagnosed with mCRPC between 01 January 2016 and 31 December 2018, who have received at least 1 line of treatment (LOT) in the mCRPC setting, and have 12 months of follow-up data available.

DETAILED DESCRIPTION:
This is a multi-country, multi-centre, retrospective, non-interventional cohort study planned to include patients diagnosed with mCRPC between 01 January 2016 and 31 December 2018, who have received at least 1 line of treatment (LOT) in the mCRPC setting, and have 12 months of follow-up data available.To describe the real-world treatment patterns in patients with mCRPC

The data will be collected retrospectively between the date of diagnosis of mCRPC (index date) and the end of follow-up, i.e., until death, the last medical record entry, or the date of data extraction, whichever is the earliest. The data on different types of treatment received by the patients, sociodemographic and clinico-pathological characteristics, and healthcare utilization will be extracted from the medical records of patients (alive or deceased) into a centrally designed electronic data capture system. For the exploratory end point on real-world treatment patterns in patients with mCSPC, data on different types of treatment received by the patients, sociodemographic and clinico-pathological characteristics will be retrospectively extracted from the medical records of patients (alive or deceased) into a centrally designed electronic data capture system.

ELIGIBILITY:
Inclusion Criteria:

* Male patients ≥18 years of age OR legal age of being an adult in the country as per local regulations 2. Patient or next of kin/legal representative (for deceased patients at study entry, unless a waiver is granted) willing and able to provide written informed consent according to the local regulations 3. Patients with a diagnosis of metastatic (stage IV) mCRPC, confirmed by either biopsy of a metastatic tumour site or by history of biopsy-proven localized disease and evidence of metastatic disease on imaging studies (which is clearly noted in hospital/clinical records) and progression on ADT alone between 01 January 2016 and 31 December 2018 4. Availability of medical records at the participating site reflecting at least one LOT received in the mCRPC setting and 12 months of follow-up from the index date (unless the patient died or was lost to follow-up within the first 12 months after diagnosis)

Exclusion Criteria:

-1. Patients with a concomitant cancer at the time of diagnosis of mCRPC or those who are treated with any anti-cancer therapy indicated for other cancers within 6 months of diagnosis of mCRPC, except for non-metastatic non-melanoma skin cancers or in situ or benign neoplasms.

2. Patients unable to give an informed consent (unless a waiver is granted)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with Metastatic Castration-resistant PROstate Cancer confirmed by pathology and/or imaging diagnosed between 01 January 2016 and 31 December 2018
Study Population: Metastatic Castration-resistant PROstate Cancer confirmed by pathology and/or imaging diagnosed
Sampling Method: Non-Probability Sample
Enrollment: 1920 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Describe the real-world treatment patterns in patients with mCRPC | 12 Months
  Proportion of patients receiving each treatment regimen for each LOT
Describe the real-world treatment patterns in patients with mCRPC | 12 Months
  Dose and DoT for each regimen for each LOT, reason(s) for stopping treatment regimen in each LOT and drug-free period D

SECONDARY OUTCOMES:
Demographic and clinico-pathological profile | 12 Months
  Describe the demographic vs clinico-pathological characteristics of patients diagnosed with mCRPC
Survival outcomes associated with different treatment regimens used for mCRPC | 12 Months
  Determine overall survival from the index date of mCRPC diagnosis
Assess the real-world effectiveness | 12 Months
  Disease progression (abstracted from clinical notes based on radiography or PSA) (including real-world progression-free survival [rwPFS] and real-world response rate [rwRR]) of different treatment regimens used for mCRPC
BRCA1/2 and HRRm status | 12 Months
  To characterize RCA1/2 and HRRm status in patients with mCRPC,

OTHER OUTCOMES:
Assess the utilization of healthcare resources during the treatment of mCRPC;(Hospitalization) | 12 Months
  Number of days of all hospitalizations and discharge with reasons for hospitalization.
Assess the utilization of healthcare resources during the treatment of mCRPC;(Healthcare Facility) | 12 Months
  Type of healthcare facility at hospitalization
Assess the utilization of healthcare resources during the treatment of mCRPC;(Insurance) | 12 Months
  Type of heath care insurance type

CONTACTS AND LOCATIONS:
Locations (24):
- Research Site, Valledupar, Colombia
- Egypt (3):
  - Research Site, Alexandria
  - Research Site, Cairo
  - Research Site, Luxor
- India (9):
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Faridabad, Haryana
  - Research Site, Srinagar, Jammu and Kashmir
  - Research Site, Bengaluru, Karnataka
  - Research Site, Mumbai, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Bhubaneshwar, Odisha
  - Research Site, Secundrabad, Telangana
  - Research Site, Howrah, West Bengal
- Research Site, Lima, Peru
- Research Site, Riyadh, Saudi Arabia
- South Korea (6):
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Gangnam-gu, Seoul
  - Research Site, Jongno-gu, Seoul
  - Research Site, Seocho-gu, Seoul
  - Research Site, Seodaemun-gu, Seoul
- Research Site, Turkey, Turkey, Turkey (Türkiye)
- United Arab Emirates (2):
  - Research Site, Alain, United Arab Emirates
  - Research Site, Dubai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Manneh R, Hashem T, Young JJ, Joshi A, Bahadir S, Omar A, Eid S, Elsayes A, Gonzalez F, Elsayed M, Kantharaju P. A REtrospective Study to Describe the Real-World Treatment Landscape in Patients with Metastatic Castration-Resistant PROstate Cancer: REMPRO. Adv Ther. 2026 Jan 12. doi: 10.1007/s12325-025-03472-5. Online ahead of print. PMID 41525044
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0817R00037&attachmentIdentifier=17ed34ca-2e15-4cdf-aa91-2a1010b133c5&fileName=REMPRO_CSR_v0.1_21Aug2023_Synopsis__Redacted.pdf&versionIdentifier=